CLINICAL TRIAL: NCT03994432
Title: Effect of Mediterranean Diet and Physical Activity in Patients With Symptomatic Endometriosis in Therapy With Estrogen-progestins or Progestins: a Randomized Controlled Trial
Brief Title: Effect of Mediterranean Diet and Physical Activity in Patients With Endometriosis
Acronym: PHAMEDENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 833_2018bis
Record Dates: First submitted 2019-03-25; First posted 2019-06-21 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis
Keywords: mediterranean diet; endometriosis; physical activity; 7 minutes work-out
MeSH Terms: conditions — Endometriosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): patients with symptomatic endometriosis in therapy with estro-progestins or progestins, who will be asked to follow a mediterranean diet and to practice an aerobic physical exercise according to the "7-minutes workout" model
  Interventions: Behavioral: intervention group
- Control group (No Intervention): patients with symptomatic endometriosis in therapy with estro-progestins or progestins.

INTERVENTIONS:
Behavioral: intervention group — follow a mediterranean diet and practice a regular aerobic exercise according to the "7-minutes workout" model.
  Arms: Intervention group

SUMMARY:
The main aim of this study is to evaluate whether a dietary recommendation based on the Mediterranean diet's principles associated with a regular aerobic physical activity, according to the "7 minutes workout", may improve pain symptoms in patients with symptomatic endometriosis (pelvic pain with numerical rating scale, NRS ≥ 4), in therapy with estrogen-progestins or progestins.

DETAILED DESCRIPTION:
Endometriosis is an estrogen-dependent inflammatory disease, affecting almost 5% of the female population during the reproductive period. The most common symptom of women with endometriosis is dysmenorrhea. Nowadays, the main therapy is pharmacological treatment (estrogen-progestins and progestins); diet and physical exercises may represent a complementary and feasible approach to reduce the pain symptoms related to this disease.

Indeed, diet may be involved in several pathophysiological mechanisms linked to endometriosis, due to its ability to influence positively or negatively prostaglandins' metabolism, chronic inflammatory processes and circulating estrogen levels.

Among the various dietary regimes, the Mediterranean diet shows many anti-inflammatory and anti-oxidant properties.

Also regular physical activity can affect positively endometriosis, due to various etiopathogenetic mechanisms including the decrease of estrogenic levels and ovulatory frequency, the increase in SHBG levels, and the modulation of cytokines in an anti-inflammatory way.

One of the reasons of low regular physical activity is the lack of free time. For this reason, the American College of Sports Medicine developed a program designed for most of the population, called "7-minutes workout". It consists in 12 high-intensity physical exercises, lasting 30 seconds each and spaced out 10 seconds of short breaks, to be performed 2-3 times a week.

Currently, there are few studies evaluating the impact of regular physical activity and Mediterranean diet regimen on endometriosis.

The objective of this randomized controlled trial is to evaluate the potential beneficial impact of regular aerobic physical activity and Mediterranean diet on endometriosis pain symptoms.

Eligible women will be selected among those attending the Endometriosis Clinic of the "L. Mangiagalli ", IRCCS Ca 'Granda Foundation and Ospedale Maggiore Policlinico, and will be randomized into two homogeneous groups ("intervention" and "control") with a 1:1 ratio, according to the type of therapy: estro-progestins or progestins.

The "intervention" group will be composed of women with symptomatic endometriosis in estro-progestins or only progestin therapy, who will be asked to follow a Mediterranean diet and to practice a regular exercise program according to the "7-minutes workout" model. The "control" group will be composed of women with symptomatic endometriosis under therapy with estro-progestins or progestins who will continue to receive the routine clinical care.

All patients participating in the study will undergo clinical and ultrasonographic evaluation every fourth months. On these occasions, women will be routinely asked to complete some questionnaires, one on pain (a numerical rating scale, NRS), one on quality of life (the Short Form-12 questionnaire, SF-12), one on psychological status (the Hospital Anxiety and Depression scale, HADS), one on sexual functioning (theFemale Sexual Function Index, FSFI) and one on the global impression of change (Patients' Global Impression of Change scale, PGIC). Women will be also asked to rate the degree of satisfaction with their treatment. Moreover, at the beginning and at the end of the study all participants will be asked to complete a dietary questionnaire, a physical activity questionnaire (International Physical Activity Questionnaire, IPAQ) and a sleep quality questionnaire (The Pittsburgh Sleep Quality Index, PSQI).

Only the patients in the "intervention" group will be asked to follow a Mediterranean diet. They will receive a nutritional counseling with the investigator's hospital dietician periodically. Furthermore, these patients will follow an aerobic physical activity program 2-3 times a week for one year.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45 years
* body mass index between 18 and 29.9
* women with symptomatic endometriosis (pelvic pain with NRS score ≥ 4), in therapy with estro-progestins or progestins
* not seeking conception

Exclusion Criteria:

* associated diseases that cause pelvic pain regardless of the presence of endometriosis, or chronic intestinal diseases (Crohn's disease or ulcerative rectocolitis).
* patients in note for all kind of surgery
* women who conduct a strong physical activity.
* women who follow vegetarian-vegan diet regimens.
* metabolic diseases that require specific dietary indications (diabetes and celiac disease, food allergies).
* medical contraindications to proposed physical activity.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Pelvic pain changes in patients with endometriosis who follow a mediterranean diet and a regular physical activity | 12 months
  The presence and severity of dysmenorrhea, deep dyspareunia, and non-menstrual pelvic pain will be assessed using an 11-point numeric rating scale (NRS), with 0 indicating absence of pain and 10 pain as bad as it could be. Scores 1 to 4 will be considered mild pain, 5 to 7 moderate pain, and 8 to 10 severe pain. Patients will be considered for enrollment if they complained of at least moderate or severe pelvic pain (NRS score ≥ 4).

SECONDARY OUTCOMES:
The degree of satisfaction in patients with endometriosis who follow a mediterranean diet and a regular physical activity | 12 months
  Patients will rate the degree of satisfaction with their treatment according to a five-category scale (very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, very dissatisfied).
Changes in state of anxiety and depression in patients with endometriosis who follow a mediterranean diet and a regular physical activity | 12 months
  To determine states of anxiety and depression we'll use the Hospital Anxiety and Depression Scale (HADS) that is a self-assessment mood scale specifically designed for use in non-psychiatric hospital outpatients. It comprises 14 questions, 7 for the anxiety subscale and 7 for the depression subscale. Lower scores indicate better psychological status.
Changes in sexual dysfunction and sexual satisfaction in patients with endometriosis who follow a mediterranean diet and a regular physical activity | 12 months
  We'll use the Female Sexual Function Index (FSFI) questionnaire that is a 19-item, multidimensional, self-report instrument for evaluating the main categories of female sexual dysfunction and sexual satisfaction. Domains include desire, arousal, lubrication, orgasm, satisfaction and pain. Each domain is scored on a scale of 1 to 5, and the maximum transformed full-scale score is 36, with a minimum full-scale score of 2.0. Women with a FSFI total score below 26.55 are categorized as experiencing sexual dysfunction
Changes in quality of life in patients with endometriosis who follow a mediterranean diet and a regular physical activity. | 12 months
  Quality of life will be assessed with the Short-Form 12 (SF-12) health survey, developed from the original SF-36 questionnaire, a well-known, validated self-administered 12-item instrument. It measures health dimensions covering functional status, well-being, and overall health. Information from the 12 items is used to construct physical (PCS-12) and mental (MCS-12) component summary measures, with higher scores indicating better health perception.
Changes in global improvement over time in patients with endometriosis who follow a mediterranean diet and a regular physical activity. | 12 months
  Overall improvement will be assessed by participants using the Patient Global Impression of Change scale, a 7-point categorical scale recommended for use in chronic pain studies as a core outcome measure of global improvement over time.According to this single-item rating system, the response during treatment is indicated by choosing one among seven alternative options, i.e., "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," and "very much worse."

CONTACTS AND LOCATIONS:
Locations (1):
- Laura Buggio Centro Endometriosi e Metrorragie Clinica Mangiagalli, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy